CLINICAL TRIAL: NCT04578223
Title: Platelet Reactivity and Treatment With Prostacyclin Analogues in Pulmonary Arterial Hypertension
Acronym: PAPAYA
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: European Health Centre Otwock (Unknown)
Responsible Party: Sponsor
Other Study IDs: KB/138/217
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Hypertension
Keywords: prostacyclin analogues; pulmonary arterial hypertension; platelet reactivity; extracellular vesicles; thrombus formation
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with pulmonary arterial hypertension treated with prostacyclin analogues on top of ERA or PDE-5i.
- Control group: Patients with pulmonary arterial hypertension treated with ERA or PDE-5i only.

SUMMARY:
Background: Prostacyclin analogues (epoprostenol, treprostinil and iloprost) induce vasodilation in advanced pulmonary arterial hypertension (PAH) but also inhibit platelets, increasing patients' bleeding risk. The antiplatelet effects of different prostacyclin analogues have never been compared head-to-head. The goal of the PAPAYA (Platelet Reactivity and Treatment With Prostacyclin Analogues in Pulmonary Arterial Hypertension) trial is(i) to compare platelet function (platelet reactivity, extracellular vesicles concentration and thrombus formation) in patients with PAH treated with prostacyclin analogues on top of endothelin receptor antagonists (ERA) and/or phosphodiesterase type 5 inhibitors (PDE5i) and patients treated only with ERA and PDE5i, and (ii) to compare the antiplatelet effect of different prostacyclin analogues.

Venous blood will be collected from patients treated with prostacyclin analogues (study group; n=40) and patients treated with ERA or PDE5i (control group; n=40). Platelet reactivity will be analysed in whole blood by impedance aggregometry using arachidonic acid, adenosine diphosphate and thrombin receptor-activating peptide as agonists. Concentrations of extracellular vesicles from all platelets (CD61+), activated platelets (CD62P+), leukocytes (CD45+) and endothelial cells (CD146+) will be analysed in platelet-depleted plasma using flow cytometry (A-60 Micro). Platelet-rich thrombus formation will be measured using whole blood perfusion system. The study will determine the antiplatelet effect of prostacyclin analogues and compare different prostacyclin analogues head-to-head to identify the best drugs to use in case of thrombosis or bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study
* Pulmonary arterial hypertension confirmed with right heart catheterization
* Treatment with prostacyclin analogues (epoprostenol, treprostinil, iloprost) - study group
* Treatment with endothelin receptor antagonists and phosphodiesterase type 5 inhibitors - control group

Exclusion Criteria:

* Known coagulopathy
* Active pathological bleeding
* Known history of bleeding disorder
* Severe thrombocytopenia (platelet count < 50,000/μL )
* Need for antiplatelet therapy with acetylsalicylic acid or P2Y12 antagonists
* Severe chronic renal failure (estimated glomerular filtration rate < 30 mL/min)
* Severe liver insufficiency (Child-Pugh class C)
* Known pregnancy, breast-feeding, or intention to become pregnant during the study period
* Study drug intolerance
* Participation in any previous study with prostacyclin analogues

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were eligible for enrolment if they (i) had PAH diagnosed according to the criteria of European Society of Cardiology and European Respiratory Society, confirmed during right heart catheterization, (ii) were treated with prostacyclin analogues on top of other drugs (study group) or only other drugs (ERA and PDE-5i; control group) for at least 1 month.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | July 5, 2017 - November 30, 2019
  Difference in platelet reactivity between patients treated with prostacyclin analogues and treated with ERA and/ or PDE5-i, assessed using impedance aggregometry

SECONDARY OUTCOMES:
Concentration of extracellular vesicles from platelets, leukocytes and endothelial cells | July 5, 2017 - November 30, 2019
  Differences in concentration of extracellular vesicles from platelets, leukocytes and endothelial cells between patients treated with prostacyclin analogues and treated with ERA and/ or PDE5i, assessed using flow cytometry
Platelet-rich thrombus formation parameters | July 5, 2017 - November 30, 2019
  Differences in platelet-rich thrombus formation parameters between patients treated with prostacyclin analogues and treated with ERA and/ or PDE5i, assessed using whole-blood flow-chamber perfusion system

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Circulation, Thromboembolic Diseases and Cardiology, Centre of Postgraduate Education Medical, European Health Centre Otwock, Warsaw, Poland